CLINICAL TRIAL: NCT06342310
Title: A Multicenter, Randomized, Double-Blind, Parallel-Group Dose-Controlled Study Evaluating the Safety and Efficacy of RE104 for Injection in the Treatment of Patients With Postpartum Depression (PPD)
Brief Title: RE104 Safety and Efficacy Study in Postpartum Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Reunion Neuroscience Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RE104-201-PPD
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-05

CONDITIONS: Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1.5 mg RE104 (Active Comparator): A single subcutaneous injection of 1.5 mg RE104 for Injection
  Interventions: Drug: RE104 for Injection
- 30 mg RE104 (Experimental): A single subcutaneous injection of 30 mg RE104 for Injection
  Interventions: Drug: RE104 for Injection

INTERVENTIONS:
Drug: RE104 for Injection — Single, subcutaneous dose of RE104 for Injection

SUMMARY:
The purpose of this study is to determine if treatment with a single dose of RE104 for Injection reduces depressive symptoms in participants with moderate-to-severe postpartum depression (PPD) as compared to active-placebo.

ELIGIBILITY:
Inclusion Criteria:

* Is ≤15 months postpartum at Screening.
* Meet DSM-5 criteria for postpartum depression (PPD): experiencing a major depressive episode that began at any time starting at the beginning of the second trimester (≥14 weeks) of pregnancy through 4 weeks post delivery.
* Has a Hamilton Depression Scale (HAM-D) total score meeting severity threshold at Screening and Baseline.
* Is not using any psychotropic medications or psychotherapy for 30 days prior to Screening, OR are on an already stable/established regimen of SSRIs or psychotherapy for 30 days prior to Screening.
* Has ceased breastfeeding at Screening.
* Has a negative pregnancy test at Screening and Day 0 prior to study drug administration.

Exclusion Criteria:

* History or active postpartum psychosis per Investigator assessment.
* History of treatment-resistant depression within the current postpartum depressive episode.
* Has a significant risk of suicide.
* Active or medical history of bipolar disorder, schizophrenia, schizoaffective disorder, psychotic disorder and/or borderline personality disorder, or first-degree family history of psychosis or bipolar disorder.
* Medically significant condition rendering unsuitability for the study .
* Has received electroconvulsive therapy (ECT) or transcranial magnetic stimulation within 90 days prior to Screening.
* Has used psychedelics such as psilocybin, ayahuasca, mescaline, or LSD (with the exception of cannabis) within 12 months prior to Screening.
* Has used or will need to use prohibited medications.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2024-06-14 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
RE104 30 mg versus RE104 1.5 mg change from baseline in MADRS total score | Day 7
  Montgomery-Åsberg Depression Rating Scale (MADRS) is a 10-item clinician rated scale measuring depression severity. The total score ranges from 0-60 with higher scores representing greater severity of depression.

SECONDARY OUTCOMES:
RE104 30 mg versus RE104 1.5 mg change from baseline in MADRS total score | Day 1, Day 14 and Day 28
  Montgomery-Åsberg Depression Rating Scale (MADRS) is a 10-item clinician rated scale measuring depression severity. The total score ranges from 0-60 with higher scores representing greater severity of depression.
RE104 30 mg versus RE104 1.5 mg percentage of patients with MADRS response (≥ 50 percent reduction in score from baseline) | Day 7
  Montgomery-Åsberg Depression Rating Scale (MADRS) is a 10-item clinician rated scale measuring depression severity. The total score ranges from 0-60 with higher scores representing greater severity of depression.
RE104 30 mg versus RE104 1.5 mg percentage of patients with MADRS remission (score ≤ to 10) | Day 7
  Montgomery-Åsberg Depression Rating Scale (MADRS) is a 10-item clinician rated scale measuring depression severity. The total score ranges from 0-60 with higher scores representing greater severity of depression.
RE104 30 mg versus RE104 1.5 mg Clinical Global Impression-Improvement (CGI-I) | Day 1, Day 7 and Day 28
  The Clinical Global Impression - Improvement (CGI-I) Scale is a clinician-rated instrument that weighs the clinical impact of the identified symptom(s) on behavior and function and measures changes in psychopathology since the treatment was administered on a scale from 1 (very much improved) to 7 (very much worse).
RE104 30 mg versus RE104 1.5 mg change from baseline in CGI-Severity (CGI-S) | Day 1, Day 7 and Day 28
  The Clinical Global Impression - Severity Scale is a clinician-rated instrument that grades severity of symptoms on a scale from 1 (normal, not ill at all) to 7 (among the most extremely ill patients).
RE104 30 mg versus RE104 1.5 mg changes in total score from baseline in Hamilton Anxiety Rating Scale (HAM-A) | Day 7
  The Hamilton Rating Scale for Anxiety (HAM-A) is a 14-item scale that is used to rate the severity of symptoms of anxiety. The total score ranges from 0-56 with higher scores representing greater severity of anxiety.
RE104 30 mg versus RE104 1.5 mg incidence of treatment-emergent adverse events (TEAEs) by frequency, severity and seriousness. | From dosing through study completion (post-dose follow-up is for 28 days)
  A treatment-emergent adverse event (TEAE) is defined as any unfavorable and unintended sign, symptom or disease temporally associated with the use of a study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Jasna Hocevar-Trnka, M.D., Study Director — Reunion Neuroscience Inc
Locations (34):
- United States (34):
  - Reunion Investigational Site, Birmingham, Alabama
  - Reunion Investigational Site, Tucson, Arizona
  - Reunion Investigational Site, Santa Monica, California
  - Reunion Investigational Site, Boulder, Colorado
  - Reunion Investigational Site, Denver, Colorado
  - Reunion Investigational Site, Lauderhill, Florida
  - Reunion Investigational Site, Tampa, Florida
  - Reunion Investigational Site, Atlanta, Georgia
  - Reunion Investigational Site, Decatur, Georgia
  - Reunion Investigational Site, Marietta, Georgia
  - Reunion Investigational Site, Savannah, Georgia
  - Reunion Investigational Site, Honolulu, Hawaii
  - Reunion Investigational Site, Kansas City, Kansas
  - Reunion Investigational Site, Shreveport, Louisiana
  - Reunion Investigational Site, Baltimore, Maryland
  - Reunion Investigational Site, Rockville, Maryland
  - Reunion Investigational Site, Springfield, Massachusetts
  - Reunion Investigational Site, Novi, Michigan
  - Reunion Investigational Site, Albuquerque, New Mexico
  - Reunion Investigational Site, Buffalo, New York
  - Reunion Investigational Site, New York, New York
  - Reunion Investigational Site, Chapel Hill, North Carolina
  - Reunion Investigational Site, Monroe, North Carolina
  - Reunion Investigational Site, Cleveland, Ohio
  - Reunion Investigational Site, Columbus, Ohio
  - Reunion Investigational Site, West Chester, Pennsylvania
  - Reunion Investigational Site, Austin, Texas
  - Reunion Investigational Site, Plano, Texas
  - Reunion Investigational Site, San Antonio, Texas
  - Reunion Investigational Site, Draper, Utah
  - Reunion Investigational Site, Salt Lake City, Utah
  - Reunion Investigational Site, Charlottesville, Virginia
  - Reunion Investigational Site, Seattle, Washington
  - Reunion Investigational Site, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No
Data sharing will be consistent with the results submission policy of ClinicalTrials.gov.